CLINICAL TRIAL: NCT07204574
Title: The Phase 1b/IIa, Open-label, Dose Escalation and Dose Expansion to Evaluate Safety, Tolerability, and Preliminary Efficacy of the Combination of HCB101, Cetuximab/Bevacizumab, and FOLFOX/FOLFIRI in Advanced or Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: FBD Biologics Limited (Industry)
Responsible Party: Principal Investigator, Hung-Chih Hsu, Attending Physician, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202401753A0
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: CRC
MeSH Terms: interventions — Bevacizumab; Cetuximab; Fluorouracil; Leucovorin; Irinotecan; Folfox protocol; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: HCB101+ Bevacizumab/Cetuximab+ Cetuximab/FOLFOX (Experimental)
  Interventions: Drug: HCB101; Drug: Bevacizumab; Drug: Cetuximab (Erbitux); Drug: FOLFIRI (Fluorouracil (5-FU), leucovorin, irinotecan); Drug: FOLFOX (Oxaliplatin/Leucovorin/5-Fluorouracil)

INTERVENTIONS:
Drug: HCB101 — QW
Drug: Bevacizumab — 5 mg/kg IV infusion, Day 1, Every 2 weeks
Drug: Cetuximab (Erbitux) — * Initial dose: 400 mg/m² IV infusion, over >2 hours, Day 1
  * Maintenance dose: 250 mg/m² IV infusion, over 60 minutes, Day 1, weekly OR 500 mg/m² IV infusion, over >2 hours, Day 1, every 2 weeks
Drug: FOLFIRI (Fluorouracil (5-FU), leucovorin, irinotecan) — Irinotecan: 180 mg/m² IV infusion over 30-90 minutes, Day 1, Every 2 weeks Folinic acid (Leucovorin): 400 mg/m² IV infusion over 2 hours, Day 1, Every 2 weeks 5-Fluorouracil (5-FU): 400 mg/m² IV bolus, Day 1; then 1200 mg/(m²·day) × 2 days continuous IV infusion (total 2400 mg/m² over 46-48 hours, Every 2 weeks
Drug: FOLFOX (Oxaliplatin/Leucovorin/5-Fluorouracil) — Folinic acid (Leucovorin): 400 mg/m² IV infusion over 2 hours, Day 1, Every 2 weeks 5-Fluorouracil (5-FU): 400 mg/m² IV bolus, Day 1; then 1200 mg/(m²·day) × 2 days continuous IV infusion (total 2400 mg/m² over 46-48 hours), Every 2 weeks Oxaliplatin: 85 mg/m² IV infusion over 2 hours, Day 1, Every 2 weeks

SUMMARY:
This is a non-randomized, open-label, dose-escalation and dose-expansion phase I/II clinical study to evaluate the safety, tolerability, and efficacy of HCB101 in combination with Cetuximab/Bevacizumab, and FOLFOX/FOLFIRI in Advanced or Metastatic Colorectal Cancer. The trial consists of two phases: the dose-escalation phase (I) and the dose-expansion phase (II).

Subjects will receive a weekly single dose of HCB101 IV infusion over 60 (±10) minutes on Days 1, 8, and 15 in each 21-day cycle in combination with Bevacizumab (5 mg/kg IV day 1; given every 14 days) /Cetuximab (500 mg/m2 IV day 1; given every 14 days) , and FOLFIRI/FOLFOX until unacceptable AE(s), radiographic or clinically documented disease progression, withdrawal of consent, loss to follow-up, death, or termination of the study whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are able to understand and willing to provide signed informed consent as described in Appendix 1, Section 10.1.3, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol, including study visits and study-related procedures.
2. Male and female subjects of ≥18 years of age, inclusive, at the time of signing the informed consent.
3. With histologically/cytologically confirmed diagnosis of unresectable locally advanced or metastatic colorectal cancer, with both RAS and BRAF wild-type, who have experienced treatment failure with prior chemotherapy for locally advanced or metastatic disease (intended for second-line treatment). Previous chemotherapy may have included 5-FU, oxaliplatin, or irinotecan.
4. Must have at least 1 measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
5. Must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at Screening.
6. Able to provide archived or fresh tumor tissue samples for CD47 expression, immune score, and whole-exome sequencing (WES) analysis, if applicable.
7. Have a life expectancy of ≥12 weeks (according to the Investigator's judgment).
8. Have adequate organ function, as indicated by the following laboratory parameters in below (had not received a blood transfusion, apheresis infusion, erythropoietin, granulocyte colony-stimulating factor, and other relevant medical support within 14 days prior to the administration of the first dose of study intervention).

   -- a) Absolute neutrophil count ≥1.5 × 109/L

   -- b) Platelets ≥75 × 109/L

   -- c) Hemoglobin ≥9.5 g/dL
   * d) Total bilirubin ≤1.5 × upper limit of normal (ULN), <3.0 × ULN if known Gilbert's disease
   * e) Alanine aminotransferase and aspartate aminotransferase ≤3× ULN and ≤5× ULN for subject with liver metastasis
   * f) Creatinine clearance ≥30 mL/min (using Cockcroft Gault equation)
   * g) Coagulation: International normalized ratio (INR), prothrombin time (PT), and activated partial thromboplastin time (aPTT) ≤1.5× ULN (The INR applies only to subjects who do not receive therapeutic anticoagulation).
9. A) Female subjects should meet at least 1 of the following criteria before they can participate in the study:

   1. Females who have no childbearing potential (i.e., physiologically incapable of pregnancy), including those who have undergone hysterectomy, bilateral oophorectomy, or bilateral salpingectomy.
   2. Postmenopausal (total cessation of menses for ≥ 1 year).
   3. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test during the Screening Period (within 7 days prior to the first dose of the study intervention), must not be lactating, and must be willing to practice a highly effective contraceptive method throughout the study (i.e., from study entry up to 6 months after the last dose of the study intervention). A highly effective method of contraception is defined as one that results in a low failure rate, i.e., less than 1% per year when used consistently and correctly. For the definition of WOCBP and highly effective methods of contraception.

B) Male subjects are eligible to participate in the study if they have undergone a vasectomy or agree to use a highly effective method of contraception and refrain from donating sperm from study entry up to 6 months after the last dose of the study intervention.

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

-Medical Conditions

1. With a known history of hypersensitivity to any components of the study intervention.
2. With other malignancies requiring treatment within 2 years prior to the first dose will be excluded, except for locally curable basal cell or squamous cell skin cancer treated with curative intent, and other malignancies with no recurrence within 2 years.
3. Primary tumor in the central nervous system (CNS), or active or untreated CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate, provided they are clinically stable for at least 28 days and have no evidence of new or enlarging brain metastases and no requirements for high-dose corticosteroids 14 days prior to dosing with study intervention. Subjects on low-dose corticosteroids (<20 mg prednisone or equivalent per day) may participate.
4. Clinically significant cardiovascular condition, including:

   • History of congestive heart failure (New York Heart Association Class >2);
   * History of unstable angina within 6 months prior to the first dose of study intervention;
   * New-onset angina or myocardial infarction within 6 months prior to the first dose of study intervention;
   * New-onset of atrial fibrillation, supraventricular arrhythmia, or ventricular arrhythmia within 6 months prior to the first dose of study intervention and still in unstable condition and requiring treatment or intervention. History of atrial fibrillation, supraventricular arrhythmia, or ventricular arrhythmia will be allowed, provided the condition is stably controlled.
5. History or presence of an abnormal ECG that, in the Investigator's opinion, is clinically meaningful (including QT interval corrected for heart rate using Fridericia's correction [QTcF] >470 msec at Screening, pacemaker installation, or previous diagnosis of congenital long QT syndrome).
6. Any previous treatment-related toxicities which have not recovered to ≤ Grade 1 as evaluated by National Cancer Institute, Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 or baseline, except alopecia and anemia (Note: subjects with chronic Grade 2 toxicities which are well managed and stable may be eligible per the discretion of the Investigator after discussion with the Sponsor and medical monitor, e.g., Grade 2 chemotherapy-induced neuropathy.)

6. With known inherited or acquired bleeding disorders or bleeding diathesis. 7. Known congenital or acquired bleeding disorders or bleeding tendency. 8. Have RBC transfusion dependence defined as requiring more than 2 units of RBC transfusions during the 4-week period prior to Screening.

9. With a previously documented diagnosis of hemolytic anemia or Evans Syndrome in the last 3 months.

Prior/Concomitant Therapy/Treatment 10. Subjects who have undergone major surgery, or have undergone radical radiotherapy within 28 days prior to the first dose of study intervention.

11. Subjects who have undergone palliative radiotherapy within 14 days prior to the first dose of study intervention,=.

12. Subjects who have used a radioactive drug (Strontium, Samarium, etc.) within 56 days prior to the first dose of the study intervention.

13. Any investigational or approved systemic cancer therapy (including chemotherapy, immunotherapy, hormonal therapy, and herbal/alternative therapies with anti-cancer indications or targeted therapy) administered within 14 days or 5 half lives, whichever is longer, prior to the first dose of the study intervention.

14. Have used herbal medication within 14 days prior to the first dose of the study intervention.

15. Active use of vitamin K antagonist anticoagulant like warfarin. Use of low molecular weight heparin and factor Xa inhibitors will be permitted on a case-by-case basis. There will be no restriction for daily aspirin ≤ 100 mg/QD.

16. Have received any treatment targeting the CD47 or SIRPα pathway. 17. Received or planning to receive live virus or bacterial vaccine within 28 days prior to the first dose of study intervention while the subject receives the study intervention. Subjects who require Corona Virus Disease 2019 (COVID-19) vaccination while on study intervention must receive a non-live vaccine (e.g., one based on messenger RNA [mRNA] or fully inactivated/genetically modified viruses incapable of replication).

Prior/Concurrent Clinical Study Experience 18. Participation in another clinical study with an investigational product administered in the last 14 days or 5 half-lives (whichever is longer) prior to receiving the first dose of study intervention. Or An investigational device was used within 28 days prior to the first dose of study intervention.

Infections 19. An uncontrolled acute infection, an active infection requiring systemic treatment, or subjects who have received systemic antibiotics within 14 days prior to the first dose of the study intervention (Note: prophylaxis use of systemic antibiotics treatment for upper tract infection is allowed as long as there is no violation of the requirement of concomitant medications).

20. Known history of human immunodeficiency virus (HIV) infection and/or acquired immunodeficiency syndrome or positive HIV testing having CD4+ T-cell counts <350 cells/µL or subjects with unknown HIV infection status who are unwilling to undergo HIV testing.

21. Known active hepatitis B or C. Subjects with hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) antibody positive test results during Screening must be further tested for hepatitis B virus (HBV) deoxyribonucleic acid (DNA) titer (excluding subjects with a DNA titer of more than 2500 copies [cps]/mL or 500 IU/mL) and HCV ribonucleic acid (RNA) (excluding subjects with an HCV RNA concentration exceeding the lower detection limit of the assay) to exclude active hepatitis B or hepatitis C infection requiring treatment. Hepatitis B virus carriers, i.e., subjects with stable hepatitis B infection after drug treatment (DNA titer not exceeding 2500 cps/mL or 500 IU/mL) and hepatitis C infected subjects who received treatment and achieved sustained virologic response for at least 12 weeks can be enrolled. Note: If the lower detection limit of the HBV DNA assay is higher than 2500 cps/mL or 500 IU/mL, the subjects with an HBV DNA assay result lower than the lower detection limit of the assay can be enrolled.

22. Active tuberculosis. 23. Known to have a history of alcoholism or drug abuse. 24. Any other medical (e.g., Child-Pugh class B or C, pulmonary, metabolic, congenital, endocrinal or CNS disease, etc.), psychiatric, or social condition deemed by the Investigator to be likely to interfere with a subject's rights, safety, welfare or ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with MTD of HCB101 in combination with Cetuximab/Bevacizumab, and FOLFOX/FOLFIRI | 2 Years
  To evaluate the safety and efficacy of HCB101 in combination with Cetuximab/Bevacizumab, and FOLFOX/FOLFIRI
Overall Rate Response (ORR) | 2 Years
  To evaluate the safety and efficacy of HCB101 in combination with Cetuximab/Bevacizumab, and FOLFOX/FOLFIRI

SECONDARY OUTCOMES:
Number/incidence and percentage of subjects with AEs, SAEs, and TEAEs | 2 Years
  To characterize the safety profiles of HCB101 in combination with Cetuximab/Bevacizumab, and FOLFOX/FOLFIRI
Progression-Free Survival (PFS) | 2 Years
  To evaluate the anti-tumor activity of HCB101 in combination with Cetuximab/Bevacizumab, and FOLFOX/FOLFIRI

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chih Hsu, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang-Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided